CLINICAL TRIAL: NCT03793959
Title: How Does a Synbiotic Supplement Affect Iron Status During Iron Repletion in Iron Depleted Female Athletes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marywood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 808959-2
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Iron-deficiency
Keywords: female athletes; iron supplementation; prebiotic; probiotic; synbiotic; serum ferritin
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: Twenty eligible athletes (baseline Hgb:12.3±0.9g/dL; sFer:18.1±9.2µg/L) were then randomized to receive either a daily synbiotic supplement (5g prebiotic fiber + 8 billion CFU probiotic B. lactis) or placebo, along with a daily Fe supplement (140 mg FeSO4/d) for 8 weeks using a double-blind design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic Supplement (Experimental): Daily synbiotic supplement (5g prebiotic fiber + 8 billion CFU probiotic B. lactis, identical to Placebo-- white powder), along with a daily Fe supplement (140 mg FeSO4/d) for 8 weeks.
  Interventions: Dietary Supplement: Synbiotic Supplement
- Placebo Supplement (Placebo Comparator): Daily placebo supplement (5g maltodextrin, identical to Experimental -- white powder), along with a daily Fe supplement (140 mg FeSO4/d) for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic Supplement
  Other Names: Regular Girl
  Arms: Synbiotic Supplement
Dietary Supplement: Placebo
  Arms: Placebo Supplement

SUMMARY:
Iron deficiency (ID) affects ~30% of female athletes, and its consequences are highly relevant to athletic performance. Poor iron (Fe) uptake remains a major factor in the development of ID. While animal studies suggest that prebiotics may improve Fe uptake, this has not been well-studied in humans. The main objective of the proposed study is to determine the effects of synbiotic supplementation on the Fe status of ID female athletes during Fe repletion.

DETAILED DESCRIPTION:
Iron deficiency (ID) affects ~30% of female athletes, and its consequences are highly relevant to athletic performance. Poor iron (Fe) uptake remains a major factor in the development of ID. While animal studies suggest that prebiotics may improve Fe uptake, this has not been well-studied in humans. The main objective of the proposed study is to determine the effects of synbiotic supplementation on the Fe status of ID female athletes during Fe repletion. At the beginning of a training season at a Division III University, the Fe status of 28 female athletes (cross-country, lacrosse, basketball, field hockey) was screened. Twenty eligible athletes (baseline Hgb:12.3±0.9g/dL; sFer:18.1±9.2µg/L) were then randomized to receive either a daily synbiotic supplement (5g prebiotic fiber + 8 billion CFU probiotic B. lactis) or placebo, along with a daily Fe supplement (140 mg FeSO4/d) for 8 weeks using a double-blind design. Fe status and body composition were assessed at baseline, mid-point and after the trial. Participants were instructed to keep daily logs of supplement intake, physical activity, GI and other symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female, >18 y of age, athlete at Marywood University, passed NCAA-required medical screening (e.g. healthy enough to participate in sport).

Exclusion Criteria:

* Current, acute, chronic illness; severe asthma; pre-existing GI disorders known to affect iron status or aggravated by iron supplementation; not pregnant or breastfeeding; clinically-diagnosed with eating disorder; consuming iron supplement within 4 weeks of screening; hemolytic anemia, excessive alcohol consumption.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 20 (Actual)
Dates: Start 2016-08-28 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Iron status | 8 weeks
  Change in serum ferritin

CONTACTS AND LOCATIONS:
Locations (1):
- Marywood University, Scranton, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] DellaValle DM, Haas JD. Iron supplementation improves energetic efficiency in iron-depleted female rowers. Med Sci Sports Exerc. 2014 Jun;46(6):1204-15. doi: 10.1249/MSS.0000000000000208. PMID 24195864
- [Background] DellaValle DM. Iron supplementation for female athletes: effects on iron status and performance outcomes. Curr Sports Med Rep. 2013 Jul-Aug;12(4):234-9. doi: 10.1249/JSR.0b013e31829a6f6b. PMID 23851410
- [Background] Dellavalle DM, Haas JD. Iron status is associated with endurance performance and training in female rowers. Med Sci Sports Exerc. 2012 Aug;44(8):1552-9. doi: 10.1249/MSS.0b013e3182517ceb. PMID 22382172
- [Background] DellaValle DM, Haas JD. Impact of iron depletion without anemia on performance in trained endurance athletes at the beginning of a training season: a study of female collegiate rowers. Int J Sport Nutr Exerc Metab. 2011 Dec;21(6):501-6. doi: 10.1123/ijsnem.21.6.501. PMID 22089308
- [Background] Laparra JM, Diez-Municio M, Herrero M, Moreno FJ. Structural differences of prebiotic oligosaccharides influence their capability to enhance iron absorption in deficient rats. Food Funct. 2014 Oct;5(10):2430-7. doi: 10.1039/c4fo00504j. Epub 2014 Aug 11. PMID 25109275